CLINICAL TRIAL: NCT03398863
Title: Intrauterine Cleaning After Delivery of Placenta During Cesarean Section
Brief Title: Intra-uterine Cleaning During Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Raghda Elsayed Ghonem, Principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dr Raghda
Record Dates: First submitted 2017-12-28; First posted 2018-01-16 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cleaning of uterine cavity (Active Comparator): Cleaning of uterine cavity: participants will have their uterine cavities cleaned with a dry laparotomy sponge after delivery of the placenta. Per standard protocol, the uterus will be explored with one hand holding a sponge to remove any remaining membranes or placental tissue, while the other hand is placed on the fundus to stabilize the uterus
  Interventions: Procedure: Cleaning of uterine cavity
- Not cleaning of uterine cavity (No Intervention): These participants will have their uterine cavities left alone after complete delivery of the placenta. The placenta will be inspected after delivery to make sure it is complete, including the membranes.

INTERVENTIONS:
Procedure: Cleaning of uterine cavity — Procedure: Cleaning the uterine cavity These participants will have their uterine cavities cleaned with a dry laparotomy sponge after delivery of the placenta. Per standard protocol, the uterus will be explored with one hand holding a sponge to remove any remaining membranes or placental tissue, while the other hand is placed on the fundus to stabilize the uterus
  Arms: Cleaning of uterine cavity

SUMMARY:
400 women who came to our Department for Cesarean Section delivery will be divided into 2 groups: Group1:Cleaning the uterine cavity "200 patients" Group2:No Cleaning of uterine cavity "200 patients"

DETAILED DESCRIPTION:
Caesarean section is the most common major surgical procedure performed in obstetric practice. The American College of Obstetricians and Gynecologists (ACOG) estimates that in 2011 alone, one in three women who gave birth in the United States did so by cesarean delivery. Compared to vaginal births, the increasing rate of caesarean births worldwide is a well known cause of maternal morbidity, including hemorrhage, anesthetic complications, shock, cardiac arrest, acute renal failure, assisted ventilation, venous thromboembolism and increased risk of major postpartum infection.

With increasing cesarean section rates and its associated complications, obstetricians are challenged to reduce perioperative and postoperative morbidity by adapting their surgical skills and techniques. Over the years, randomized clinical trials have tried to answer many questions surrounding the safety of several cesarean section techniques that impart maternal morbidity. For example, the optimal type of cesarean section skin incision, whether or not to create a bladder flap, one layer versus two later closure of the uterus, irrigating the abdominal cavity, closure versus non closure of the parietal peritoneum, and suture versus staples for skin closure at cesarean section.

Cleaning the uterine cavity following cesarean section is a routine practice by many obstetricians. To ensure that the entire placenta and membranes are removed after delivery of the placenta at cesarean, the uterine cavity is usually cleaned with one hand holding a dry sponge to remove any remaining membranes or placental tissue, while the other hand is placed on the fundus to stabilize the uterus. However, despite the lack of evidence to support a policy of routine intrauterine cleaning after placental delivery at cesarean section, the benefits of intrauterine cleaning as a routine practice during cesarean sections remains uncertain. Obstetricians who do not routinely clean the uterine cavity after placental delivery argue that this procedure is not performed routinely after vaginal deliveries, and thus is a justification not to do so during cesarean sections

ELIGIBILITY:
Inclusion Criteria:

* women age from 20 to35 years old with intact membrane women with singleton or multiple pregnancy women with cephalic or breech presentation

Exclusion Criteria:

* premature rupture of membranes chorioamnionitis Diabetes mellitus Immunosuppressive disorder or therapy Fetal demise

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Postpartum endometritis | Within weeks
  Endomyometritis after delivery [ Time Frame: Within 6 weeks after delivery ] Endomyometritis will be diagnosed by the presence of two or more of the following: abnormally tender uterus on examination, temperature more than 38.0°C at any time postoperatively, and unexplained maternal tachycardia more than 100 beats per minute (bpm). A diagnosis of endomyometritis will be criteria for initiating treatment with antibiotics.
  Endomyometritis after delivery [ Time Frame: Within 6 weeks after delivery ] Endomyometritis will be diagnosed by the presence of two or more of the following: abnormally tender uterus on examination, temperature more than 38.0°C at any time postoperatively, and unexplained maternal tachycardia more than 100 beats per minute (bpm). A diagnosis of endomyometritis will be criteria for initiating treatment with antibiotics.

SECONDARY OUTCOMES:
Primary postpartum hemorrhage | Within 6 weeks
  Post partum hemorrhage [ Time Frame: Within 6 weeks after delivery ] Mean surgical time [ Time Frame: Immediately post cesarean ]
  Calculated blood loss [ Time Frame: Within 6 weeks post delivery ] Hospital length of stay [ Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 4 days postpartum ] Return of gastrointestinal function [ Time Frame: Participants will be followed for the duration to return of bowel function, an expected average of 2 days postpartum ] Repeat surgery [ Time Frame: Within 6 weeks post delivery ] Hospital readmission rates. [ Time Frame: Within 6 weeks post delivery ]

CONTACTS AND LOCATIONS:
Overall Officials: Dr yasser Abou talib, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Ain shams University, Cairo
  - Faculty of Medicine-Ainshams University, Cairo